CLINICAL TRIAL: NCT04940650
Title: Detection of Myocardial Inflammation in Cyclists After Strenuous Exercise: a Pilot Study Part 1
Brief Title: COUREUR Study Myocardial Inflammation in Cyclist Part 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021/020
Record Dates: First submitted 2021-06-18; First posted 2021-06-25 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Myocardial Inflammation
MeSH Terms: conditions — Myocarditis | interventions — Exercise Test; Echocardiography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recreational cyclists performing the 'étape du tour (EDT) de France 2021 (Other)
  Interventions: Diagnostic Test: exercise testing; Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: exercise testing — To define the strenuous physical exercise in this study, each participant will be asked to perform two hours of high intensity (HIT)-effort during the endurance exercise of at least 6 to 7 hours. Therefore all participants will have exercise testing approximately 1 week before the physical exercise to set aerobic and anaerobic gas exchange thresholds, as well as VO2max.
Diagnostic Test: Echocardiography — Measurements of mass, volumes and function will be obtained of both the left and right ventricles at rest enabling comparisons with cardiac MRI and traditional echo measures.

SUMMARY:
The study will evaluate myocardial inflammation in cyclists after high intense and sustained exercise. Our hypothesis is that strenuous exercise in recreational cyclists may be associated with myocardial inflammation. Myocardial fibrosis in asymptomatic athletes is associated with life-threatening arrhythmic events and sudden death. Although myocarditis seems to be the most likely underlying cause, it remains unclear if strenuous and sustained physical exercise can cause myocardial inflammation with development of myocyte necrosis and possibly myocardial fibrosis in athletes.

Nineteen recreational cyclists performing "L'ETAPE DU TOUR (EDT) de France" a cycling ride (175 km, 3600 m of positive altitude difference) on July 4 2021 will be included in this study.

In part 1 of the study, each participant will complete a detailed questionnaire detailing their training history and an echocardiography at rest will be performed. All participants will have exercise testing approximately 1 week before the EDT stage to set aerobic and anaerobic gas exchange thresholds, as well as VO2max.

ELIGIBILITY:
Inclusion Criteria:

* Recreational cyclists performing the 'étape du tour (EDT) de France 2021 ride

Exclusion Criteria:

* presence of pre-existing cardiovascular or pulmonary diseases, hypertension, diabetes, peripheral vascular diseases, any inflammatory or auto-immune diseases and the intake of anti-inflammatory drugs.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
DETECTION OF MYOCARDIAL INFLAMMATION IN CYCLISTS AFTER STRENUOUS EXERCISE: A PILOT STUDY PART 1 | approximately 1 week before the strenuous exercise
  Aerobic and anaerobic gas exchange heart rate thresholds, and VO2max (ml/kg/min) will be measured in all cyclists approximately 1 week before the high intense exercise. This exercise testing will be performed to evaluate high-intensity exercise as factor of exercise-induced myocardial inflammation in cyclists.
DETECTION OF MYOCARDIAL INFLAMMATION IN CYCLISTS AFTER STRENUOUS EXERCISE: A PILOT STUDY PART 1 | approximately 1 week before the strenuous exercise
  Assessments of weight (in kilograms) and heigth (in meters) to determine VO2 max (ml/kg/min)

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Hasselt University, Hasselt
  - Jessa Hospital, Hasselt

REFERENCES:
- [Derived] Ghekiere O, Herbots L, Peters B, Berg BV, Dresselaers T, Franssen W, Padovani B, Ducreux D, Ferrari E, Nchimi A, Demanez S, De Bosscher R, Willems R, Heidbuchel H, La Gerche A, Claessen G, Bogaert J, Eijnde BO. Exercise-induced myocardial T1 increase and right ventricular dysfunction in recreational cyclists: a CMR study. Eur J Appl Physiol. 2023 Oct;123(10):2107-2117. doi: 10.1007/s00421-023-05259-4. Epub 2023 Jul 22. PMID 37480391